CLINICAL TRIAL: NCT01871246
Title: Acute Exacerbation of COPD and Physical Activity - Preliminary Study
Status: Terminated | Type: Observational
Why Stopped: The study was not funded and we ran out of resources to complete the data analysis. This was a qualitative study and requires substantial time and effort to conduct data analysis.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Janet L. Larson, Professor, University of Michigan
Other Study IDs: HUM00062912
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- People with COPD & recent exacerbation: The group consists of people with COPD who have had an exacerbation in the last year.

SUMMARY:
People with chronic obstructive pulmonary disease (COPD) are very sedentary and efforts to establish an active lifestyle are challenging because of periodic acute exacerbations of COPD that interrupt physical activity patterns and contribute to further decline in physical activity. The purpose of this preliminary research is to learn more about the experience of acute exacerbations of COPD (AECOPD) from the perspective of the patient and his/her family and to learn how AECOPDs affect physical activity.

DETAILED DESCRIPTION:
Individuals with chronic obstructive pulmonary disease (COPD) are very sedentary and their physical activity is often interrupted by acute exacerbations of COPD (AECOPD). Little is known about the expectations had by individuals with COPD and the effects of these expectations on their physical activity. To increase the understanding of these expectations in people with COPD, a study is proposed to explore their experience of daily fluctuations in symptoms and AECOPDs, focusing on how these experiences influence health promoting behaviors, especially physical activity (PA).

This study will involve an enrollment visit during which consent will be obtained, survey data will be administered (that they may take home), spirometry testing will be conducted, and a physical activity monitor (ActivPAL device) will be applied to be worn one week to allow us to understand their usual PA. A clinical ethnographic interview will then be conducted one week following enrollment, at which point the questionnaires and ActivPAL device will be collected. A second clinical ethnographic interview will be conducted one week following the first. Survey data will again collected at week 15 by mail.

ELIGIBILITY:
Inclusion Criteria:

* People who have emphysema or chronic bronchitis as their primary health problem
* People who have had a respiratory infection or an exacerbation of their COPD within the last year.
* People who are 55 years or older
* Family member of someone who meets the above criteria.

Exclusion Criteria:

* Other lung diseases as their primary pulmonary problem.
* Mobility problems that limit physical activity

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with COPD, who have had an exaccerbation in the last year who live in the greater Ann Arbor area and their family members.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Physical activity during AECOPD | week 1
  Subjects will be asked to report how they managed their physical activity during the last AECOPD. Current physical activity will be measured with accelerometry and by the CHAMPS questionnaire.

SECONDARY OUTCOMES:
Sense of coherence | week 1 and week 15
  Questionnaire that measures one's global orientation to life and the extent to which one sees life as comprehensible, manageable and meaningful.
Barriers efficacy scale | week 1 week 15
  Questionnaire that measures barriers to exercise and physical activity. The subjects reports the level of confidence they have that they can overcome each barrier.
Help seeking behavior | week 1 and week 15
  Questionnaire assesses help seeking with respect to healthcare services.
COPD Stigma Scale | week 1 and week 15
  Questionnaire measures the stigma associated with having COPD.

OTHER OUTCOMES:
Social Support for Exercise | week 1
  Questionnaire measures social support, positive and negative social influences for physical activity and social support for exercise.
COPD symptoms | week 1
  Questionnaire, the COPD Assessment Tests quantifies severity of the most recent exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Larson, PhD, Principal Investigator — University of Michigan - School of Nursing
Locations (1):
- University of Michigan - School of Nursing, Ann Arbor, Michigan, United States